CLINICAL TRIAL: NCT05594615
Title: A NON-RANDOMIZED, MULTIPLE-DOSE, OPEN-LABEL, SINGLE SEQUENCE STUDY TO EVALUATE THE EFFECT OF CONCOMITANT ADMINISTRATION OF EDP-235 ON THE PHARMACOKINETICS AND SAFETY OF MIDAZOLAM, CAFFEINE, AND ROSUVASTATIN IN HEALTHY PARTICIPANTS
Brief Title: Drug-Drug Interaction Study Between EDP-235, Midazolam, Caffeine and Rosuvastatin in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Enanta Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EDP 235-003
Record Dates: First submitted 2022-10-21; First posted 2022-10-26 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: COVID-19
Keywords: drug-drug interaction
MeSH Terms: conditions — COVID-19 | interventions — EDP-235; Midazolam; Rosuvastatin Calcium; Caffeine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- EDP-235, midazolam, rosuvastatin and caffeine (Experimental): Subjects will receive EDP-235, midazolam, rosuvastatin and caffeine throughout the treatment period on respective dosing days
  Interventions: Drug: EDP-235; Drug: Midazolam; Drug: Rosuvastatin; Drug: Caffeine

INTERVENTIONS:
Drug: EDP-235 — Subjects will receive EDP-235 once daily on Days 5-15
Drug: Midazolam — Subjects will receive midazolam once daily on Days 1 and 12
Drug: Rosuvastatin — Subjects will receive rosuvastatin once daily on Days 2 and 13
Drug: Caffeine — Subjects will receive caffeine once daily on Days 1 and 12

SUMMARY:
A Drug-Drug Interaction study to assess the effects of EDP-235 on the Pharmacokinetics and Safety of midazolam, caffeine and rosuvastatin.

ELIGIBILITY:
Inclusion Criteria:

* An informed consent document signed and dated by the subject
* Healthy male and female subjects of any ethnic origin between the ages of 18 and 55 years, inclusive
* Screening body mass index (BMI) of 18 to 30 kg/m2 with a minimum body weight of 50 kg
* Female subjects of childbearing potential must agree to use two effective methods of contraception from the date of Screening until 90 days after the last dose of EDP-235. A male participant who has not had a vasectomy and is sexually active with a woman of childbearing potential must agree to use effective contraception from the date of Screening to 90 days after his last dose of study drug.

Exclusion Criteria:

* Clinically relevant evidence or history of illness or disease
* Pregnant or nursing females
* History of febrile illness within 7 days prior to the first dose of study drug or subjects with evidence of active infection
* A positive urine drug screen at Screening or Day -1
* Current tobacco smokers or use of tobacco within 3 months prior to Screening.
* Any condition possibly affecting drug absorption (e.g., gastrectomy, cholecystectomy)
* History of regular alcohol consumption
* Participation in a clinical trial within 30 days prior to the first dose of study drug
* History of drug allergy to midazolam, caffeine, or rosuvastatin

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2022-10-06 (Actual); Primary Completion 2022-11-04 (Actual); Study Completion 2022-11-18 (Actual)

PRIMARY OUTCOMES:
Cmax of midazolam, caffeine, and rosuvastatin with and without the coadministration of EDP-235 | Up to 17 Days
AUC of midazolam, caffeine, and rosuvastatin with and without the coadministration of EDP-235 | Up to 17 Days

SECONDARY OUTCOMES:
Safety measured by adverse events | Up to 22 days

CONTACTS AND LOCATIONS:
Overall Officials: Enanta Pharmaceuticals, Inc, Study Director — Enanta Pharmaceuticals, Inc
Locations (1):
- ICON, plc., Salt Lake City, Utah, United States